CLINICAL TRIAL: NCT02611622
Title: Impact of Multimedia-based Patient Education on Patient Satisfaction Scores in an Otolaryngology Practice Setting
Brief Title: LumaENT and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201301163
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Control (Active Comparator): * Participants will be presented with envelopes labeled with a unique block-randomization code and asked to pick one
  * Once the participant selects an envelope, the research coordinator will verify whether the code assigns the patient to the control or the intervention group, without the knowledge of the otolaryngologist who will be blinded to participant randomization at this point.
  * Participants in the control group will proceed to filling out Demographic Survey and Patient Satisfaction Survey
  * Once completed, they will be given the opportunity to discuss any further questions or concerns about their thyroid condition with their otolaryngologist
  Interventions: Other: Survey
- Arm 2: LUMA ENT™ (Experimental): * Participants will be presented with envelopes labeled with a unique block-randomization code and asked to pick one
  * Once the participant selects an envelope, the research coordinator will verify whether the code assigns the patient to the control or the intervention group, without the knowledge of the otolaryngologist who will be blinded to participant randomization at this point.
  * Participants in the intervention group will proceed to viewing the LUMA ENT™ videos pertinent to their thyroid condition using either of the two iPADS (the videos should not last longer than 10 minutes)
  * Once video viewing is complete, participants will be given the opportunity to discuss any further questions or concerns about their thyroid condition with their otolaryngologist, especially as relates to questions that arise as a result of viewing the video
  * Subsequently, the participants will proceed to filling out Demographic Survey and Patient Satisfaction Survey
  Interventions: Behavioral: LUMA ENT™; Other: Survey

INTERVENTIONS:
Behavioral: LUMA ENT™
  Arms: Arm 2: LUMA ENT™
Other: Survey — Demographic and Patient Satisfaction Survey

SUMMARY:
Patient satisfaction is an important metric currently used to rate quality of healthcare in hospitals. Maximizing patient satisfaction scores is therefore significantly beneficial to any hospital establishment. Recent studies have shown patient satisfaction depends on multiple factors, including patient involvement in treatment decision-making processes and patients' knowledge of treatment options. Internal review of departmental patient satisfaction survey scores revealed deficits in the aforementioned areas of patient satisfaction, with the domains of "how well concerns were addressed", "explanation of tests and procedures" and "effort to include patients in decisions" having the lowest scores on patient satisfaction surveys. This highlights the gap in patient satisfaction that the Otolaryngology department seeks to improve on, so as to maximize patient satisfaction, and in turn, the quality of healthcare provided.

The aim of this study is to assess the improvement in patient satisfaction scores that can be obtained by incorporating LUMA ENT™, a disease-specific multimedia patient education software, into the treatment decisions for thyroid disorders. LUMA ENT™ is a leading patient education software that provides visual anatomic animations of disease processes, disease progression and treatment options to improve patients' knowledge. Thyroid disorders have been chosen for study due to their high frequency of occurrence in the patient population and generalizability to a wide medical audience.

The investigators will perform a single-blinded randomized-controlled study of patients visiting the physician practices of the Department of Otolaryngology for management of thyroid disorders. Participants will be randomized into control and intervention groups. Upon completion of the routine physician-patient clinical encounter, the intervention group will view a 5- minute LUMA ENT™ video discussing their specific thyroid condition, its natural progression history, and treatment options. They will have an opportunity to ask the physician any further questions that arise from viewing the video. The control group will not view the LUMA ENT video. Patient satisfaction surveys will then be provided to both groups at the end of the visit as is routinely done and scores subsequently compared.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients scheduled to visit the BJH/WU Department of Otolaryngology clinic for management of thyroid disorders (ranging from benign to cancerous nodules or masses) that will involve surgical interventions of complete or partial thyroidectomies.
* must be between the ages of 18 and 80
* may be male or female
* must understand spoken or written English language
* must be able to provide informed consent

Exclusion Criteria:

-Patients who have already undergone any thyroid surgery will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-08-07 (Actual); Primary Completion 2015-10-21 (Actual); Study Completion 2015-10-21 (Actual)

PRIMARY OUTCOMES:
Evaluate improvement in patient satisfaction scores obtained with the incorporation of LUMA ENT™ in pre-treatment counseling | Day 1
  To compare survey domain scores, MANOVA will be used to explore differences between groups and control for confounders.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Nussenbaum, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu